CLINICAL TRIAL: NCT03889509
Title: A Systematic Review of Factors Associated With Pulmonary Arterial Hypertension in Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Janet Pope, Professor of Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: YJJEP0001
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Arterial Hypertension; Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; pulmonary hypertension; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Scleroderma, Systemic; Scleroderma, Diffuse; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol is of a systematic review for risk factors of pulmonary arterial hypertension in systemic sclerosis.

DETAILED DESCRIPTION:
A systematic review was conducted to determine the risk/associated factors for pulmonary arterial hypertension in systemic sclerosis, including clinical/disease characteristics, antibody status, test results and biomarkers. The frequency of publications featuring a risk/association were reported. The following databases were searched: Medline, EMBASE, the Cochrane Library, Web of Science, and SCOPUS.

The following search terms were used:

( essential pulmonary hypertension or familial primary pulmonary hypertension or hypertension, pulmonary or hypertension,lung or hypertensive pulmonary vascular disease or idiopathic pulmonary arterial hypertension or lung arterial hypertension or lung artery hypertension or lung hypertension or primary pulmonary hypertension or pulmonary arterial hypertension or pulmonary artery hypertension or pulmonary fixed hypertension or pulmonary hypertensive disease or pulmonary hypertensive diseases or pulmonary hypertensive disorder or pulmonary hypertensive disorders )

AND

( generalised scleroderma or generalized scleroderma or progressive scleroderma or progressive sclerodermia or progressive sclerosis,systemic or progressive systemic sclerosis or scleroderma, generalised or scleroderma, generalized or scleroderma, progressive or scleroderma, systemic or sclerosis,progressive systemic or sclerosis,systemic or sclerosis,systemic progressive or systemic progressive sclerosis or systemic scleroderma or systemic sclerosis,progressive or

scleroderma, limited or limited scleroderma or limited cutaneous scleroderma or

diffuse scleroderma or progressive diffuse scleroderma or scleroderma, diffuse )

AND

( prevalence or prevalence study or relative risk or risk factors )

ELIGIBILITY:
Inclusion Criteria:

* Studies were included they were (1) in patients with SSc; and if they (2) determined PAH with right heart catheterization; (3) involved a comparison of SSc patients with and without PAH; and (4) had sample size larger than 20.

Exclusion Criteria:

* Studies were excluded if they were review articles, and if the study was written in languages other than English. When the same patients were used in more than one analysis, the most recent or largest sample-size study was included.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study reflects a search strategy of available literature on pulmonary arterial hypertension in scleroderma.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Pulmonary arterial hypertension in scleroderma | 2 years from study start date
  to determine the prevalence associated with pulmonary arterial hypertension in scleroderma
Risk factors for pulmonary arterial hypertension in scleroderma | 2 years from study start date
  to determine the risk factors associated with pulmonary arterial hypertension in scleroderma

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD MPH, Principal Investigator — St. Joseph's healthcare London
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada